CLINICAL TRIAL: NCT01559506
Title: ABS to Reduce Contamination in Spine Surgery
Brief Title: Air Barrier System Device to Reduce Contamination in Posterior Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nimbic Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ABS-003
Record Dates: First submitted 2012-03-14; First posted 2012-03-21 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Surgery
Keywords: CFU; surgery site

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No device (No Intervention): Subject does not receive ABS system
- Air Barrier System device (Experimental): Device is deployed adjacent to the surgery site and activated.
  Interventions: Device: Air Barrier System device

INTERVENTIONS:
Device: Air Barrier System device — Device is deployed adjacent to the surgery site and activated.
  Arms: Air Barrier System device

SUMMARY:
The objective of this study is to determine whether the Air Barrier System (ABS) reduces airborne colony-forming units (e.g. bacteria) present at surgery sites during posterior spinal procedures

DETAILED DESCRIPTION:
The ABS is a device that uses localized clean air flow to shield a surgery site from ambient airborne contamination. This study examines the hypothesis that the ABS can reduce the presence of airborne colony-forming units at the surgery site during posterior spinal procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing lumbar and cervical laminectomy with instrumentation.

Exclusion Criteria:

* Active infection
* Prior prosthesis infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih O Darouiche, MD, Principal Investigator — Baylor College of Medicine; Sean Self, Principal Investigator — Nimbic Systems
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Device | Air Barrier System Device
Started | 20 | 21
Completed | 20 | 18
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Device | Air Barrier System Device | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: CFU Density
Description: Colony-forming unit density at incision site (CFU/m3)
Time Frame: Surgical case CFU density will be determined at up to 1 month from completion of surgical cases
Measure: Mean (95% Confidence Interval); unit: CFU/m^3
Arm/Group | No Device | Air Barrier System Device
Number analyzed (Participants) | 20 | 18
CFU/m^3 | 5.05 [2.45 to 7.65] | 1.55 [1.08 to 2.01]

ADVERSE EVENTS:
Arm/Group | No Device | Air Barrier System Device
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No